CLINICAL TRIAL: NCT00969150
Title: A Double-blind, Placebo-Controlled, Flexible-Dose Study of F2695 SR in Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of Levomilnacipran ER (F2695 SR) in Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LVM-MD-02
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-08

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Levomilnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Matching placebo capsules, oral administration, once daily dosing.
  Interventions: Drug: Placebo
- 1 (Experimental): Levomilnacipran ER capsules, flexible dose, oral administration, once daily dosing.
  Interventions: Drug: Levomilnacipran ER

INTERVENTIONS:
Drug: Levomilnacipran ER — Drug: Levomilnacipran ER (flexible dose) Study drug is to be given orally, in capsule form, once daily, for 8 weeks.
  Arms: 1
Drug: Placebo — Matching placebo to be given orally, in capsule form, once daily, for 8 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of Levomilnacipran ER versus placebo in the treatment of outpatients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-80 years old
* Currently meet the DSM-IV-TR criteria for Major Depressive Disorder
* The patient's current depressive episode must be at least 4 weeks in duration

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women with childbearing potential who are not practicing a reliable method of birth control
* Patients with a history of meeting DSM-IV-TR criteria for:

  * any manic or hypomanic episode
  * schizophrenia or any other psychotic disorder
  * obsessive-compulsive disorder
* Patients who are considered a suicide risk

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Gommoll, MS, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Locations (24):
- United States (24):
  - Forest Investigative Site, Scottsdale, Arizona
  - Forest Investigative Site, Encino, California
  - Forest Investigative Site, Los Alamitos, California
  - Forest Investigative Site, Oceanside, California
  - Forest Investigative Site, Denver, Colorado
  - Forest Investigative Site, Jacksonville, Florida
  - Forest Investigative Site, Orlando, Florida
  - Forest Investigative Site, Chicago, Illinois
  - Forest Investigative Site, Wichita, Kansas
  - Forest Investigative Site, Glen Burnie, Maryland
  - Forest Investigative Site, Fall River, Massachusetts
  - Forest Investigative Site, East Lansing, Michigan
  - Forest Investigative Site, Cherry Hill, New Jersey
  - Forest Investigative Site, Brooklyn, New York
  - Forest Investigative Site, New York, New York
  - Forest Investigative Site, Staten Island, New York
  - Forest Investigative Site 013, Canton, Ohio
  - Forest Investigative Site, Dayton, Ohio
  - Forest Investigative Site, Portland, Oregon
  - Forest Investigative Site, Philadelphia, Pennsylvania
  - Forest Investigative Site, Lincoln, Rhode Island
  - Forest Investigative Site, Woodstock, Vermont
  - Forest Investigative Site, Bellevue, Washington
  - Forest Investigative Site, Seattle, Washington

REFERENCES:
- [Derived] Gommoll CP, Greenberg WM, Chen C. A randomized, double-blind, placebo-controlled study of flexible doses of levomilnacipran ER (40-120 mg/day) in patients with major depressive disorder. J Drug Assess. 2014 Jan 16;3(1):10-9. doi: 10.3109/21556660.2014.884505. eCollection 2014. PMID 27536449
- [Derived] Cutler AJ, Gommoll CP, Chen C, Greenberg WM, Ruth A. Levomilnacipran Extended-Release Treatment in Patients With Major Depressive Disorder: Improvements in Functional Impairment Categories. Prim Care Companion CNS Disord. 2015 Jun 11;17(3):10.4088/PCC.14m01753. doi: 10.4088/PCC.14m01753. eCollection 2015. PMID 26644957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited over a 12-month period from September of 2009 to September of 2010 at 24 studies sites in the United States.
Pre-assignment Details: Patients went through a 1-week single-blind placebo run-in period immediately preceding an 8-week double-blind treatment period.
Groups:
- Placebo: Dose Matched placebo capsules, oral administration, once daily dosing for 8 weeks.
- Levomilnacipran ER: Levomilnacipran ER capsules, flexible dose, oral administration, once daily dosing for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Levomilnacipran ER
Started | 182 | 175
Completed | 149 | 135
Not Completed | 33 | 40
Not completed — Adverse Event | 4 | 14
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 9 | 12
Not completed — Withdrawal by Subject | 13 | 9
Not completed — Lost to Follow-up | 5 | 4
Not completed — Other reasons | 1 | 0

BASELINE CHARACTERISTICS:
Population: While a total of 362 patients were randomized to receive double-blind treatment, 5 of these patients were either lost to follow up or withdrew consent before receiving double-blind treatment. The Baseline Participant population is based on the 357 randomized patients who went on to receive double-blind treatment (Safety Population).
Groups:
- Placebo: Matching placebo capsules, oral administration, once daily dosing for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Levomilnacipran ER | Total
Number analyzed (Participants) | 182 | 175 | 357
Age Continuous [Mean (Standard Deviation); unit: years] | 43.7 (13.3) | 42.8 (12.9) | 43.3 (13.1)
Age, Customized [Number; unit: participants]
  18 years to 19 years | 2 | 1 | 3
  20 years to 29 years | 33 | 34 | 67
  30 years to 39 years | 35 | 32 | 67
  40 years to 49 years | 47 | 53 | 100
  50 years to 59 years | 40 | 37 | 77
  60 years to 80 years | 25 | 18 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 99 | 215
  Male | 66 | 76 | 142
Race/Ethnicity, Customized [Number; unit: participants]
  White | 149 | 133 | 282
  Black or African American | 28 | 29 | 57
  Asian | 3 | 4 | 7
  American Indian or Alaska native | 0 | 3 | 3
  Other | 2 | 6 | 8
  Hispanic or Latino | 18 | 16 | 34
  Not Hispanic or Latino | 164 | 159 | 323
Region of Enrollment [Number; unit: participants]
  United States | 182 | 175 | 357
Weight [Mean (Standard Deviation); unit: kg] | 82.9 (18.0) | 82.4 (18.1) | 82.7 (18.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms Per Meter Squared] | 28.9 (5.7) | 28.7 (5.4) | 28.8 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: MADRS was used to assess depressive symptomatology during the past week. Patients are rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest.
  Each item of the 10 items are scored on a 7-point scale. A score of 0 indicates the absence of symptoms,and a score of 6 indicates symptoms of maximum severity. The total MADRS score for this measure ranges from 0 (absence of symptoms) to 60 (maximum severity).
Time Frame: From Baseline to Week 8
Population: Of the 357 patients who received at least 1 dose of double-blind treatment (Safety Population), 355 patients had at least 1 postbaseline MADRS assessment (Intent to Treat [ITT] Population).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Levomilnacipran ER
Number analyzed (Participants) | 181 | 174
units on a scale | -14.2 (0.90) | -15.7 (0.94)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran ER; Test type: Superiority or Other; p = 0.2492, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -1.49, 95% CI 2-sided [-4.02 to 1.05]

2. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale (SDS) is a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point continuum (0 = no impairment to 10 = most severe) with the total SDS score ranging from 0 (no impairment) to 30 (most severe)
Time Frame: From Baseline to Week 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Levomilnacipran ER
Number analyzed (Participants) | 181 | 174
units on a scale | -8.2 (0.67) | -8.8 (0.68)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran ER; Test type: Superiority or Other; p = 0.5625, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -0.54, 95% CI 2-sided [-2.38 to 1.29]

ADVERSE EVENTS:
Time Frame: Adverse event data was collection over a 14-month period from September 2009 to November 2010 at 24 study sites in the U.S.
Description: The Serious Adverse Event data presented here is for the safety population. The Other Adverse Event data presented here is for the safety population during the 8 week double-blind treatment period.
Arm/Group | Placebo | Levomilnacipran ER
Serious Adverse Events (participants affected / at risk) | 1/182 | 0/175
Other Adverse Events (participants affected / at risk) | 58/182 | 90/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=182) | Levomilnacipran ER (N=175)
Blood Pressure Increased (Investigations) | 1 | 0
Chest Pain (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=182) | Levomilnacipran ER (N=175)
Nausea (Gastrointestinal disorders) | 6 | 30
Headache (Nervous system disorders) | 22 | 28
Dry mouth (Gastrointestinal disorders) | 11 | 14
Ejaculation disorder (Reproductive system and breast disorders) | 0/66 | 6/76
Insomnia (Psychiatric disorders) | 13 | 12
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 12
Dizziness (Nervous system disorders) | 3 | 11
Upper respiratory tract infection (Infections and infestations) | 11 | 6
Vomiting (Gastrointestinal disorders) | 1 | 10
Erectile dysfunction (Reproductive system and breast disorders) | 1/66 | 4/76
Heart rate increased (Investigations) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.